CLINICAL TRIAL: NCT00121069
Title: Placebo-Controlled Pilot Study of Escitalopram in the Treatment of Specific Phobia
Brief Title: Study of Escitalopram in the Treatment of Specific Phobia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Connor, Kathryn M., M.D. (Individual)
Collaborators: Forest Laboratories (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3990-02-9
Record Dates: First submitted 2005-07-13; First posted 2005-07-21 (Estimated); Last update posted 2005-07-21 (Estimated); Status verified 2005-07

CONDITIONS: Phobic Disorders
Keywords: specific phobia; anxiety; SSRI; clinical trial; escitalopram
MeSH Terms: conditions — Phobic Disorders; Phobia, Specific; Anxiety Disorders | interventions — Escitalopram

INTERVENTIONS:
Drug: Escitalopram

SUMMARY:
This pilot study is designed to assess the efficacy of escitalopram in the treatment of specific phobia in adult outpatients.

DETAILED DESCRIPTION:
This double-blind placebo-controlled pilot trial study is designed to assess the efficacy of 12 weeks of escitalopram vs. placebo in the treatment of specific phobia in adult outpatients. It is hypothesized that escitalopram is safe and effective in the treatment of specific phobia.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65 years of age
* DSM-IV criteria for specific phobia according to the MINI
* For women of childbearing potential, a negative serum pregnancy test at screening
* Written informed consent

Exclusion Criteria:

* Any current primary DSM-IV diagnosis other than specific phobia
* History of DSM-IV substance abuse or dependence within the last months
* Lifetime history of bipolar I disorder, schizophrenia or other psychotic disorder, mental retardation, or other pervasive developmental disorder or cognitive disorder due to a general medical condition
* Suicide risk or serious suicide attempt within the last year
* Clinically significant laboratory or EKG abnormality or unstable medical condition
* For women of childbearing potential, unwillingness to use an acceptable form of contraception during the study
* Subjects needing concurrent use of psychotropic medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2002-09; Study Completion 2004-09

PRIMARY OUTCOMES:
Response based on a criterion of 50% or greater reduction in the Marks Main Phobia Questionnaire and Marks Fear Questionnaire from baseline

SECONDARY OUTCOMES:
Response based on CGI-I category

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn M. Connor, M.D., Principal Investigator — Duke University
Locations (1):
- Dept of Psychiatry and Behvaioral Science, Duke Unviersity Medical Center, Durham, North Carolina, United States